CLINICAL TRIAL: NCT00727727
Title: Stabilization on, or Change-Over to the Non-Ergot Dopamine Agonist Piribedil in Patients With Morbus Parkinson - a Post Marketing Surveillance Study in Private Practices.
Brief Title: SEDPARK2: Post Marketing Surveillance to Observe Safety and Efficacy of Piribedil in Parkinson's Disease (PIR-002/K)
Status: Completed | Type: Observational
Sponsor: Desitin Arzneimittel GmbH (Industry)
Responsible Party: Dr. Martina Wangemann, Desitin Arzneimittel GmbH
Other Study IDs: PIR-002/K
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Parkinson's Disease
Keywords: Piribedil (trade name: Clarium); non-ergot dopamine agonist; Morbus Parkinson; Tolerability; Efficacy; Post Marketing Surveillance
MeSH Terms: conditions — Parkinson Disease | interventions — Piribedil

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parkinsonian patients
  Interventions: Drug: Piribedil

INTERVENTIONS:
Drug: Piribedil

SUMMARY:
The objective of the Post Marketing Surveillance Study is to investigate the use of the non-ergot dopamine agonist piribedil (trade name: CLARIUM) in mono- and combination therapy in patients with Morbus Parkinson. Neurologists in private practices in Germany should document the safety and course of the disease/change of parkinsonian symptoms during stabilisation on, or change over from other dopamine agonist treatment under routine conditions. Piribedil should be prescribed according to its marketing authorisation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years and older.
* Indication: Morbus Parkinson.
* Treatment with piribedil for the first time.
* Monotherapy with piribedil.
* Combination therapy with L-Dopa (from the beginning or secondary in combination with other antiparkinsonian drugs).

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Morbus Parkinson who require therapy with dopamine agonists
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
to monitor use in daily routine practice including adverse events | 3 months

SECONDARY OUTCOMES:
to monitor use in daily routine practice including efficacy aspects | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Medical Practice for Neurology, Dresden
  - Medical Practice for Neurology, Wedel

REFERENCES:
- [Background] Castro-Caldas A, Delwaide P, Jost W, Merello M, Williams A, Lamberti P, Aguilar M, Del Signore S, Cesaro P; Parkinson-Control Study Group. The Parkinson-Control study: a 1-year randomized, double-blind trial comparing piribedil (150 mg/day) with bromocriptine (25 mg/day) in early combination with levodopa in Parkinson's disease. Mov Disord. 2006 Apr;21(4):500-9. doi: 10.1002/mds.20750. PMID 16267842
- [Background] Rascol O, Dubois B, Caldas AC, Senn S, Del Signore S, Lees A; Parkinson REGAIN Study Group. Early piribedil monotherapy of Parkinson's disease: A planned seven-month report of the REGAIN study. Mov Disord. 2006 Dec;21(12):2110-5. doi: 10.1002/mds.21122. PMID 17013922
- [Background] Rascol O, Pathak A, Bagheri H, Montastruc JL. Dopaminagonists and fibrotic valvular heart disease: further considerations. Mov Disord. 2004 Dec;19(12):1524-5. doi: 10.1002/mds.20328. No abstract available. PMID 15515031